CLINICAL TRIAL: NCT00242684
Title: Manifestations, Causes, and Consequences of PEU in Elderly TCU Residents
Brief Title: PEU in Elderly TCU Residents
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: IIR 04-298
Record Dates: First submitted 2005-10-18; First posted 2005-10-20 (Estimated); Results first posted 2014-12-02 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2014-09

CONDITIONS: Aging
Keywords: Aging; Undernutrition; Inflammation; Frail Elderly
MeSH Terms: conditions — Malnutrition; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and plasma samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: older patients admitted to a TCU unit

SUMMARY:
Background: There is tremendous controversy regarding the adequacy/effectiveness of the nutritional care provided in VA Transitional Care Units (TCUs). The interrelationship between concurrent inflammatory disease, the adequacy of a resident's nutrient consumption, the development or resolution of putative nutritional deficits, and clinical outcomes is not established. Given the known obstacles to increasing nutrient intake (e.g. cost, resident acceptance, associated morbidity) and the lack of proven effectiveness of all forms of nutrition support and nutritional supplementation to improve clinical outcomes, a better understanding of these interrelationships is needed and will be the focus of this study.

Objectives: The primary objective of this study is to determine how best to define nutritional risk (i.e., risk for adverse clinical outcomes due to inadequate nutrient intake) among older VA TCU residents. As part of this objective, we will seek to develop a better understanding of the interrelationship between nutrient intake, weight change, serum concentration of albumins, health status/illness severity, and mortality. The secondary objective is to develop a prediction model for identifying which TCU residents are likely to have ongoing problems with low nutrient intake. The ultimate objective is to develop a clinically useful system to identify residents who are likely to benefit from specific interventions aimed at improving nutritional risk.

DETAILED DESCRIPTION:
Background: There is tremendous controversy regarding the adequacy/effectiveness of the nutritional care provided in VA Transitional Care Units (TCUs). The interrelationship between concurrent inflammatory disease, the adequacy of a resident's nutrient consumption, the development or resolution of putative nutritional deficits, and clinical outcomes is not established. Given the known obstacles to increasing nutrient intake (e.g. cost, resident acceptance, associated morbidity) and the lack of proven effectiveness of all forms of nutrition support and nutritional supplementation to improve clinical outcomes, a better understanding of these interrelationships is needed and will be the focus of this study.

Objectives: The primary objective of this study is to determine how best to define nutritional risk (i.e., risk for adverse clinical outcomes due to inadequate nutrient intake) among older VA TCU residents. As part of this objective, we will seek to develop a better understanding of the interrelationship between nutrient intake, weight change, serum concentration of albumins, health status/illness severity, and mortality. The secondary objective is to develop a prediction model for identifying which TCU residents are likely to have ongoing problems with low nutrient intake. The ultimate objective is to develop a clinically useful system to identify residents who are likely to benefit from specific interventions aimed at improving nutritional risk.

Methods: To meet these objectives, 400 older, non-terminally ill veterans admitted to a VA TCU (where average length of stay is approximately 90 days) will be prospectively studied using the same methodologic approach validated in prior VA hospital-based investigations. After completing a comprehensive admission assessment, each subject will be monitored closely throughout his/her TCU stay with serial nutrient intake and recurring metabolic, functional, neuropsychological, cognitive, nutritional, and medical assessments. Weights, anthropometrics, and blood for serum proteins, inflammatory markers (e.g., cytokines), and other select lab indices will be obtained at least monthly until discharged. Resting metabolic rate (by indirect calorimetry) will be obtained on select residents. Each subject will remain in the study for 12 months. From discharge through the end of the subject's study year, each subject will be monitored by phone to determine survival and days of institutional (e.g., hospital, NH) care. At study's end, strengths of associations will be assessed using univariable and multivariable analytic techniques including logistic and Cox Proportional-Hazards analyses.

Findings: See citations linked.

Status: Status: Funding began 9-1-2005. Subject recruitment began 3-1-2006. To date, we have recruited 446 subjects into the study. 446 subjects have been discharged from the inpatient phase of the study. The average length of stay for these subjects is 32 days.

Impact: Our study will provide a clearer understanding of what factors contribute to the apparent nutritional deficits seen in many older veterans residing in VA nursing home TCUs. The study will also lead to the development of a clinically useful system to identify TCU residents who are likely to benefit from specific interventions aimed at improving nutritional risk and thus clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

> 64 years of age, admitted to the TCU

Exclusion Criteria:

If they: have a terminal disease (eg end-stage organ failure refractory to medical management receiving palliate care).

Min Age: 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: non-terminally ill adults admitted to the TCU
Sampling Method: Probability Sample
Enrollment: 446 (Actual)
Dates: Start 2006-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis H. Sullivan, MD, Principal Investigator — Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR
Locations (1):
- Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR, No. Little Rock, Arkansas, United States

REFERENCES:
- [Result] Sullivan DH, Johnson LE, Dennis RA, Roberson PK, Garner KK, Padala PR, Padala KP, Bopp MM. Nutrient intake, peripheral edema, and weight change in elderly recuperative care patients. J Gerontol A Biol Sci Med Sci. 2013 Jun;68(6):712-8. doi: 10.1093/gerona/gls234. Epub 2012 Nov 26. PMID 23183900
- [Result] Dennis RA, Johnson LE, Roberson PK, Heif M, Bopp MM, Garner KK, Padala KP, Padala PR, Dubbert PM, Sullivan DH. Changes in activities of daily living, nutrient intake, and systemic inflammation in elderly adults receiving recuperative care. J Am Geriatr Soc. 2012 Dec;60(12):2246-53. doi: 10.1111/jgs.12007. Epub 2012 Nov 23. PMID 23176675
- [Result] Sullivan DH, Roberson PK, Johnson LE, Mendiratta P, Bopp MM, Bishara O. Association between inflammation-associated cytokines, serum albumins, and mortality in the elderly. J Am Med Dir Assoc. 2007 Sep;8(7):458-63. doi: 10.1016/j.jamda.2007.04.004. Epub 2007 Aug 13. PMID 17845949
- [Result] Sullivan DH, Johnson LE, Dennis RA, Roberson PK, Heif M, Garner KK, Bopp MM. The Interrelationships among albumin, nutrient intake, and inflammation in elderly recuperative care patients. J Nutr Health Aging. 2011 Apr;15(4):311-5. doi: 10.1007/s12603-010-0297-1. PMID 21437564
- [Result] Dennis RA, Johnson LE, Roberson PK, Heif M, Bopp MM, Cook J, Sullivan DH. Changes in prealbumin, nutrient intake, and systemic inflammation in elderly recuperative care patients. J Am Geriatr Soc. 2008 Jul;56(7):1270-5. doi: 10.1111/j.1532-5415.2008.01789.x. Epub 2008 Jun 10. PMID 18547360

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 540 study eligible patients admitted to the TCU between March 2006 and March 2011, 446 (83%) entered the study.
Groups:
- Transitional Care Unit Veterans: older patients admitted to a TCU unit
Period: Overall Study
Arm/Group | Transitional Care Unit Veterans
Started | 446
Completed | 446
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Elderly patients admitted to TCU
Arm/Group | Transitional Care Unit Veterans
Number analyzed (Participants) | 446
Age, Continuous [Mean (Standard Deviation); unit: Years] | 78.6 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 437
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 446
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 54
  White | 392
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Average Daily Nutrient Intake <70% of Predicted Needs
Time Frame: While hospitalized on TCU, for up to 40 days
Measure: Number; unit: percentage of subjects
Arm/Group | Transitional Care Unit Veterans
Number analyzed (Participants) | 446
percentage of subjects | 26

2. Post Hoc Outcome: Percentage of Subjects With Average Daily Nutrient Intake <90% of Predicted Needs
Time Frame: While hospitalized on TCU, for up to 40 days
Measure: Number; unit: percentage of subjects
Arm/Group | Transitional Care Unit Veterans
Number analyzed (Participants) | 446
percentage of subjects | 49

ADVERSE EVENTS:
Time Frame: Not applicable as this was an observational study
Arm/Group | Transitional Care Unit Veterans
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
This was an observational study designed to develop a better understanding of the interrelationships among nutrient intake, weight change, serum concentration of albumins, illness severity, and mortality. For more details, see cited references.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes